CLINICAL TRIAL: NCT02709681
Title: Hydroxyurea in Sickle Cell Disease: a Large Nation-wide Cohort Study From Italy
Brief Title: Hydroxyurea in the Treatment of Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Società Italiana Talassemie ed Emoglobinopatie (Other)
Responsible Party: Sponsor
Other Study IDs: SocietaITE
Record Dates: First submitted 2016-03-01; First posted 2016-03-16 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-03

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SCD patients: Patients followed in 32 Italian Centers.
  Interventions: Other: Physician standard-of-care in SCD patients

INTERVENTIONS:
Other: Physician standard-of-care in SCD patients

SUMMARY:
This is a retrospective cohort study of Sickle Cell Disease (SCD) patients attending 32 treatment centers across Italy. The aim of this study will be to report the Italian experience with the use of hydroxyurea in a large cohort of SCD patients and to evaluate the benefits and safety of this intervention for the prevention and management of a wide range of clinical morbidities

DETAILED DESCRIPTION:
The indication for hydroxyurea initiation was 2-3 vaso-occlusive crisis and/or hospitalizations in the last year.

The study will analyze demographics (age and gender), origin, genotype, clinical phenotype (vaso-occlusive or hemolytic), transfusion history (including exchange), and folic acid use, average laboratory values up to three years pre-hydroxyurea and for the period post-hydroxyurea therapy including total hemoglobin level, fetal hemoglobin level, hemoglobin S level, white blood count, platelet count, lactate dehydrogenase level, total and direct bilirubin levels, aspartate and alanine aminotransferase levels, and serum creatinine level.

The incidence of complications pre- and post-hydroxyurea therapy will be also analyzed including: stroke, silent cerebral infraction, acute chest syndrome, vaso-occlusive crisis, hospitalization, pulmonary hypertension, leg ulcers, bone necrosis, and kidney injury. Safety data included adverse events as reported by the treating physician and the incidence of malignancy or death as well as pregnancy incidents and their outcomes will be also pointed out.

ELIGIBILITY:
Inclusion Criteria:

* Sickle Cell Disease affected patients
* 2-3 vaso-occlusive crisis and/or hospitalizations in the last year

Exclusion Criteria

* none

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A population of SCD (Homozigous HbS and Beta Thal /HbS) patients followed in 32 Italian Centers was included in this analysis.
Sampling Method: Non-Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Changes in laboratory parameters is being assessed | An average of 3 years before and an average of 3 years after initiation of hydroxyurea therapy
  Increases or decreases in percentage of total hemoglobin, fetal hemoglobin and hemoglobin S level will be assessed. Changing of white blood cells and platelets counts, lactate dehydrogenase, bilirubin, aspartate aminotransferase and serum creatinine level will be also evaluated.
Changes in complication rates is being assessed | An average of 3 years before and an average of 3 years after initiation of hydroxyurea therapy
  Changing in the incidence of stroke, silent cerebral infraction, acute chest syndrome, vaso-occlusive crisis, pulmonary hypertension, leg ulcers, bone necrosis and kidney injury will be evaluated.
Rate of hospitalizations | An average of 3 years before and an average of 3 years after initiation of hydroxyurea therapy
  Changing in rate of hospitalizations before and after start hydroxyurea therapy

SECONDARY OUTCOMES:
Changing in the incidence of complications according to specific subgroups | An average of 3 years before and an average of 3 years after initiation of hydroxyurea therapy
  We also stratified the analysis according to age (≥18 years), origin (Italian and African), genotype (βS/β0, βS/β+ and βS/βS) duration of hydroxyurea treatment (≥10 years) and hydroxyurea dose(≥15 mg/kg/day).

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Rigano, MD, Principal Investigator — Servico Integrado de Tecnicas Endovasculares
Locations (30):
- Italy (30):
  - Ospedali Civili Riuniti di Sciacca, Sciacca, Agrigento
  - Ospedale Vittorio Emanuele III, Gela, Caltanisetta
  - Azienda Ospedaliero-Universitaria, Bari
  - U.O. Oncoematologia Pediatrica Ospedali Civili, Brescia
  - Ospedale "A. Perrino", Brindisi
  - Azienda Ospedaliera Universitaria Di Cagliari, Cagliari
  - Ospedale Vittorio Emanuele, Catania
  - ARNAS "Garibaldi", Catania
  - University of Catania, Catania
  - A.O. "Pugliese-Ciaccio", Catanzaro
  - Osp.San Giovanni Di Dio, Crotone
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - E.O. Ospedali Galliera, Genova
  - Università degli Studi di Milano, Milan
  - Azienda Ospedaliero-Universitaria di Modena - Policlinico, Modena
  - Clinica pediatrica Monza S. Gerardo, Monza
  - Azienda Ospedaliera San Gerardo di Monza, Monza
  - Aorn A. Cardarelli, Napoli
  - Clinica di Onco-Ematologia Pediatrica, Università di Padova, Padua
  - A.R.N.A.S. "Civico", Palermo
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Policlinico San Matteo, Pavia
  - Centro Emofilia e Medicina Trasfusionale - Pres. Ospedaliero, Ravenna
  - A. O. Bianchi Melacrino Morelli, Reggio Calabria
  - Ospedale S. Eugenio - FF UOSD DH Talassemici, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A.Gemelli, Roma
  - U.O.S. Talassemia P.O. Umberto I°, Syracuse
  - Università degli Suidi di Torino, Torino
  - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rigano P, De Franceschi L, Sainati L, Piga A, Piel FB, Cappellini MD, Fidone C, Masera N, Palazzi G, Gianesin B, Forni GL; Italian Multicenter Study of Hydroxyurea in Sickle Cell Anemia Investigators. Real-life experience with hydroxyurea in sickle cell disease: A multicenter study in a cohort of patients with heterogeneous descent. Blood Cells Mol Dis. 2018 Mar;69:82-89. doi: 10.1016/j.bcmd.2017.08.017. Epub 2017 Oct 9. PMID 29107441